CLINICAL TRIAL: NCT02166749
Title: Ultra Long-term Follow-up of the Outcome After Subtotal Versus Total Abdominal Hysterectomy
Brief Title: Clinical Follow up After Subtotal and Total Hysterectomy
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Seija Ala-Nissilä, MD, Turku University Hospital
Other Study IDs: ETMK:41/180/2010
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Abdominal Hysterectomy (& Wertheim)
Keywords: Hysterectomy, long term follow up, subjective outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subtotal abdominal hysterectomy: 107 women
  Interventions: Procedure: Subtotal abdominal hysterectomy
- Total abdominal hysterectomy: 105 women
  Interventions: Procedure: Subtotal abdominal hysterectomy

INTERVENTIONS:
Procedure: Subtotal abdominal hysterectomy — Comparison of women undergoing subtotal abdominal hysterectomy (n=107) and women with total abdominal hysterectomy (n=105) a mean of 33 years ago.
  Other Names: Total abdominal hysterectomy

SUMMARY:
The purpose of this study was to find out subjective and objective outcomes of patients undergoing subtotal or total abdominal hysterectomy during a follow up of a mean 33 years after the operation. The hypothesis is that there are similar outcomes after both types of operations.

DETAILED DESCRIPTION:
Objective: To evaluate ultra long-term follow-up after subtotal and total hysterectomy in patients operated on during 1978-1979 in Turku University Hospital, Finland.

Methods: From the original cohort of 212 patients 193 were sent a postal questionnaire in 1997 to find out possible symptoms related to hysterectomy. Again in 2011 a questionnaire based evaluation with a possibility of a clinical visit to study hospital was done for 153 patients. In the first evaluation a self-made questionnaire and in the second evaluation validated questionnaires were used. During a follow-up visit a clinical examination using also POP-Q-system was done. Additionally, hospital records of the patients were reviewed to find out subsequent operations after hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* benign indication for hysterectomy

Exclusion Criteria:

* abnormal Pap smear

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population included 212 patients operated on during February 1978 and May 1979 in Turku University Hospital. 107 women underwent subtotal and 105 women total abdominal hysterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 1997-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of participants having subjective symptoms after hysterectomy | 19 years and 33 years postoperatively
  Urinary and bowel symptoms assessed with questionnaires and Visual Analog Scale.
  Sexual symptoms assessed with questionnaire.

SECONDARY OUTCOMES:
Objective evaluation of pelvic organ prolapse after hysterectomy | 33 years postoperatively
  Gynecological examination and measurements using pelvic organ prolapse quantification system (POP-Q) to find out the number of participants having prolapse.

CONTACTS AND LOCATIONS:
Overall Officials: Juha Mäkinen, Professor, Study Director — Turku University Hospital
Locations (1):
- Department of Obstetrics and Gynecology, Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Ala-Nissila S, Haarala M, Jarvenpaa T, Makinen J. Long-term follow-up of the outcome of supracervical versus total abdominal hysterectomy. Int Urogynecol J. 2017 Feb;28(2):299-306. doi: 10.1007/s00192-016-3143-0. Epub 2016 Sep 17. PMID 27640066